CLINICAL TRIAL: NCT05061745
Title: Neuromodulation for Dysphoria
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Florida State University (Other)
Responsible Party: Principal Investigator, F. Andrew Kozel, Principal Investigator, Florida State University
Allocation: Non-Randomized | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: STUDY00002372
Record Dates: First submitted 2021-08-30; First posted 2021-09-30 (Actual); Last update posted 2026-01-22 (Actual); Status verified 2026-01

CONDITIONS: Dysphoria
Keywords: Neuromodulation

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: No

ARMS (3):
- Guided Meditation VR for Wellness (Active Comparator): Selected modules of commercially available meditation VR
  Interventions: Device: Guided Meditation VR for Wellness
- Accelerated Transcranial Magnetic Stimulation: Treatment A (Active Comparator): Intermittent theta-burst over dlPFC
  Interventions: Device: Accelerated Transcranial Magnetic Stimulation: Treatment A
- Accelerated Transcranial Magnetic Stimulation: Treatment B (Active Comparator): Intermittent theta-primed 10Hz over mPFC
  Interventions: Device: Accelerated Transcranial Magnetic Stimulation: Treatment B

INTERVENTIONS:
Device: Guided Meditation VR for Wellness — Selected Modules of Commercially Available "Guided Meditation VR" presented on Valve Index Headset
  Arms: Guided Meditation VR for Wellness
Device: Accelerated Transcranial Magnetic Stimulation: Treatment A — Either MagVenture Transcranial Magnetic Stimulation (Treatment Coil Cool B70 AP) or The NeuroStar® System will be used.
  Arms: Accelerated Transcranial Magnetic Stimulation: Treatment A
Device: Accelerated Transcranial Magnetic Stimulation: Treatment B — Either MagVenture Transcranial Magnetic Stimulation (Cool D-B80 AP) or The NeuroStar® System will be used.
  Arms: Accelerated Transcranial Magnetic Stimulation: Treatment B

SUMMARY:
This is an open label prospective pilot study of two neuromodulation interventions for patients suffering from dysphoria. Dysphoria is a transdiagnostic symptom of unease or dissatisfaction experienced across a range of diagnoses, including mood disorders and pain. There is a significant gap of treatment options across conditions with dysphoria, particularly non-medicated and self-care alternatives.

Many neuromodulation therapies require extensive medical resources or time to deliver. Thus, the investigators will test two non-invasive technologies administered in a manner that would reduce resources and/or time. Virtual Reality (VR) overlays the sensory system to block the external environment and provide vast range of meaningful sensory experiences. Transcranial Magnetic Stimulation (TMS) involves a magnetic pulse passing through the scalp to depolarize neurons in the outer cortex of the brain, and daily treatments over 6 weeks are currently FDA indicated for the treatment of major depressive disorder. Accelerated TMS is the delivery of treatment in a shorter period of time.

The primary objective of this study to demonstrate the preliminary effectiveness, tolerability, and feasibility of these two interventions: Guided Meditation VR for Wellness and Accelerated Transcranial Magnetic Stimulation.

ELIGIBILITY:
Inclusion Criteria for Arm 1:

1. Adults age 18 years and above
2. Reported symptoms of dysphoria: PHQ-9 ≥ 10; GAD-7 ≥ 10; PCL-5 ≥ 45 or Average Pain Intensity ≥ 4/10 for > 3 months - this will ensure at least moderate level of reported difficulty with mood, anxiety, trauma, or pain
3. No changes in psychotropic medication (if taking psychotropic medication) and/or supportive psychotherapy for 1 month prior to baseline visit; and clinically appropriate to maintain stable treatment regimen for duration of trial.
4. Clinically competent to give informed written consent and ability to understand study procedures and to comply with them for the entire length of the study

Exclusion Criteria for Arm 1:

1. Significant auditory or visual impairment that prevents participants from using Virtual Reality headset.
2. Neurologic conditions or devices impacting brain circuitry (e.g., ferrous metal in head, seizure disorder, brain tumor, stroke, aneurysm, multiple sclerosis, etc.)
3. Active substance use disorder or hallucinogen use in last 3 months or any current substance use that puts the participant at increased risk or significant impairment
4. Dementia or other cognitive disorder making unable to engage in treatment
5. Any history or diagnosis of Schizophrenia, Schizoaffective Disorder, Delusional Disorder or other psychotic illness that precludes safe participation in trial.
6. Suicidal risk that precludes safe participation defined as clinical impression that the participant is at significant risk for suicide.
7. OCD cannot be the primary disorder but can have OCD symptoms
8. Inability to stop taking any medication that significantly increases cortical excitability (e.g., tricyclic antidepressants, stimulants, clozapine, etc.)
9. Unstable medical conditions or any current medical condition that could preclude being able to safely participate in this phase of the study (e.g., unstable metabolic abnormality, unstable angina, etc.)
10. Severe Traumatic Brain Injury
11. We will exclude non-English speakers because of the need for rapid communication before and during the use of technology.
12. Significant ongoing litigation or claims that impact research activities, as determined by the research study team. (Research may especially be impacted when mental health or pain is being evaluated for litigation or claims, such as civil and criminal cases, disability claims and worker's compensation).
13. The following groups will NOT be included.

    * Adults unable to consent
    * Individuals who are not yet adults (infants, children, teenagers)
    * Prisoners

Inclusion for Arms 2 and 3:

1. Adults age 18 years and above
2. Reported symptom of dysphoria: PHQ-9 ≥ 10; GAD-7 ≥ 10; PCL-5 ≥ 45 or Average Pain ≥ 4/10 for > 3 months - this will ensure at least moderate level of reported difficulty with mood, anxiety, trauma, or pain
3. No changes in psychotropic medication (if taking psychotropic medication) and/or changes in supportive psychotherapy for 1 month prior to initial visit; and clinically appropriate to maintain stable treatment regimen for duration of trial
4. Clinically competent to give informed written consent and ability to understand study procedures and to comply with them for the entire length of the study

Exclusion for Arms 2 and 3 :

1. Medical contraindication for neuromodulation (e.g., ferrous metal in head, seizure disorder, brain tumor, stroke, aneurysm, multiple sclerosis, etc.)
2. Active substance use disorder in last 3 months or any current substance use that puts the participant at increased risk or significant impairment
3. Dementia or other cognitive disorder making unable to engage in treatment
4. Any history or diagnosis of Schizophrenia, Schizoaffective Disorder, delusional Disorder or other psychotic illness that precludes safe participation in trial
5. Suicidal risk that precludes safe participation defined as clinical impression that the participant is at significant risk for suicide
6. OCD cannot be the primary disorder but can have OCD symptoms
7. Inability to stop taking any medication that significantly lowers the seizure threshold (e.g., tricyclic antidepressants, clozapine, etc.)
8. Current, planned, or suspected pregnancy
9. Unstable medical conditions or any current medical condition that could preclude being able to safely participate in TMS treatment (e.g., unstable metabolic abnormality, unstable angina, etc.)
10. Severe Traumatic Brain Injury
11. We will exclude non-English speakers because of the need for rapid communication during the delivery of treatments
12. Significant ongoing litigation or claims that impact research activities, as determined by the research study team. (Research may especially be impacted when mental health or pain is being evaluated for litigation or claims, such as civil and criminal cases, disability claims and worker's compensation).
13. The following groups will NOT be included.

    * Adults unable to consent
    * Individuals who are not yet adults (infants, children, teenagers)
    * Pregnant women
    * Prisoners

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 100 (Estimated)
Dates: Start 2021-09-29 (Actual); Primary Completion 2026-08 (Estimated); Study Completion 2027-08 (Estimated)

PRIMARY OUTCOMES:
Arm 1 Hypothesis 1 | Week 2
  Primary Outcome will be determined by descriptive feasibility metrics. Feasibility will be determined by number of patients enrolled.
Arm 1 Hypothesis 2 | Week 2
  Primary Outcome measure is SF-36 Short Form for all patients.
Arm 1 Hypothesis 3 | Week 2
  Primary Outcome measure is the clinician-administered scale that tracks the designated primary disorder.
Arm 1 Hypothesis 4 | From Baseline over 10 weeks
  Primary Outcome measure is the clinician-administered scale that tracks the designated primary disorder.
Arm 2 Hypothesis 1 | Week 2
  Primary Outcome measure is the SF-36 Short Form for all participants.
Arm 2 Hypothesis 2 | Week 2
  Primary Outcome measure is the clinician-administered scale that tracks the designated primary disorder.
Arm 2-3 Hypothesis 3 | From Baseline to Week 6
  Primary Outcome measure is SF-36 Short Form for all participants.
Arm 2-3 Hypothesis 4 | Week 2
  Primary outcome (Treatments A and B). Tolerability will be assessed by side effect profile.
Arm 2-3 Hypothesis 4-Treatment B | Treatment B-Week 6
  Primary outcome (Treatments A and B). Tolerability will be assessed by side effect profile.
Arm 3 Hypothesis 5 | Treatment B - Week 2
  Primary Outcome measure is the SF-36 Short Form for all participants. Significantly greater improvement in rating scores from baseline of Treatment A Exit Visit ("Follow Up A1" or "Follow Up A5") to "Follow Up B1" will be tested (t-test).

CONTACTS AND LOCATIONS:
Overall Officials: F. Andrew Kozel, M.D., M.S.C.R., D.F.A.P.A., Principal Investigator — Florida State University
Locations (1):
- Florida State University, Tallahassee, Florida, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Senda MC, Johnson KA, Taylor IM, Jensen MM, Hou Y, Kozel FA. A Pilot Trial of Stepwise Implementation of Virtual Reality Mindfulness and Accelerated Transcranial Magnetic Stimulation Treatments for Dysphoria in Neuropsychiatric Disorders. Depress Anxiety. 2023 Nov 22;2023:9025984. doi: 10.1155/2023/9025984. eCollection 2023. PMID 40224597
- [Derived] Spitz AM, Senda MC, Johnson KA, Taylor IM, Jensen MM, Kozel FA. The Relationship of Anxious Arousal With Treatment of Dysphoria Using Virtual Reality Mindfulness and 2 Accelerated Transcranial Magnetic Stimulation Protocols. J Clin Psychiatry. 2024 May 22;85(2):23m15195. doi: 10.4088/JCP.23m15195. PMID 38780528